CLINICAL TRIAL: NCT05160363
Title: A Randomised, Double-blind, Placebo Controlled, Parallel Group Study in Healthy Adult Volunteers to Determine the Tolerability and Safety of Pyronaridine (PYR) Co-administered With Piperaquine (PQP) Under Fasted Conditions
Brief Title: A Healthy Volunteer Safety Study of Pyronaridine Tetraphosphate Taken in Combination With Piperaquine Tetraphosphate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Richmond Pharmacology Limited (Industry); PharmaKinetic Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: MMV_SMC_21_01
Record Dates: First submitted 2021-12-03; First posted 2021-12-16 (Actual); Results first posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2023-12

CONDITIONS: Healthy
MeSH Terms: interventions — pyronaridine; piperaquine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PYR and PQP Combination (Experimental): Single dose in the morning on Days 1, 2 and 3 of the study Pyronaridine tetraphosphate 540 mg (three tablets) if body weight 50kg - <65kg; OR, 720 mg (4 tablets) if body weight is ≥65 kg Piperaquine tetraphosphate 960 mg (three tablets) if body weight 50kg - <75kg; OR, 1280 mg (4 tablets) if body weight ≥75kg
  Interventions: Drug: Pyronaridine Tetraphosphate; Drug: Piperaquine tetraphosphate
- PYR and Placebo Combination (Placebo Comparator): Single dose in the morning on Days 1, 2 and 3 of the study Pyronaridine tetraphosphate 540 mg (three tablets) if body weight 50kg - <65kg; OR, 720 mg (4 tablets) if body weight is ≥65 kg Matched placebo for piperaquine (3 or 4 tablets based on body weight)
  Interventions: Drug: Pyronaridine Tetraphosphate; Drug: Placebo
- PQP and Placebo Combination (Placebo Comparator): Single dose in the morning on Days 1, 2 and 3 of the study Piperaquine tetraphosphate 960 mg (three tablets) if body weight 50kg - <75kg; OR, 1280 mg (4 tablets) if body weight ≥75kg Matched placebo for pyronaridine (3 or 4 tablets based on body weight)
  Interventions: Drug: Piperaquine tetraphosphate; Drug: Placebo
- Placebo Combination (Sham Comparator): Single dose in the morning on Days 1, 2 and 3 of the study Matched placebo for pyronaridine (3 or 4 tablets dependent on body weight) and matched placebo piperaquine (3 or 4 tablets dependent on body weight)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pyronaridine Tetraphosphate — A total of 24 participants will be dosed with pyronaridine tetraphosphate, sixteen participants will be additionally be dosed with piperaquine tetraphosphate, eight patients will additionally be dosed with placebo.
  Arms: PYR and PQP Combination; PYR and Placebo Combination
Drug: Piperaquine tetraphosphate — A total of 24 participants will be dosed with piperaquine tetraphosphate, sixteen participants will be additionally be dosed with pyronaridine tetraphosphate, eight patients will additionally be dosed with placebo.
  Arms: PQP and Placebo Combination; PYR and PQP Combination
Drug: Placebo — Placebo tablets will be administered in combination with pyronaridine tetraphosphate (8 patients), OR, in combination with piperaquine tetraphosphate (8 patients), OR, only matched placebo tablets will be administered (8 patients)
  Arms: PQP and Placebo Combination; PYR and Placebo Combination; Placebo Combination

SUMMARY:
The study is a clinical trial involving two medicines called piperaquine (PQP) and pyronaridine (PYR) which, in combination with dihydroartemisinin (DHA) and with artesunate (ART) respectively, have been in clinical use for over 20 years to treat acute episodes of malaria. PYR and PQP are both known to be well tolerated and provide effective treatment for malarial infection when administered in their licensed combinations, but have not been administered together in combination before.

This new combination is being considered for development for malaria prevention (i.e. chemoprophylaxis) in sub-Saharan Africa and therefore, the trial participants will be exclusively drawn from a population from that origin.

DETAILED DESCRIPTION:
In 2019, an estimated 229 million cases of malaria occurred worldwide, with approximately 94 % occurring in WHO African Region, leading to 409 000 deaths, of which about two thirds were in children under five years of age. In addition, there were an estimated 33 million pregnancies in the moderate to high transmission countries of the WHO African Region, of which 35 % (12 million) were exposed to malaria infection during pregnancy.

Case management with highly effective antimalarial drugs has contributed to the decrease in malaria morbidity and mortality. However, preventive administration of antimalarial drugs is also recommended for use in selected high-risk populations, irrespective of malaria infection status, both to treat any unrecognized Plasmodium infections and to prevent new ones. These preventive treatments prevent or cure undetected malarial illness with the goal to achieve therapeutic drug levels in the blood throughout the period of greatest risk (WHO 2021). WHO strongly recommends with a high-certainty evidence the following malaria chemopreventive therapies: seasonal malaria chemoprevention (SMC), intermittent preventive treatment in infants (IPTi), and intermittent preventive treatment of malaria in pregnancy (IPTp).

Despite the strong public health evidence of chemoprevention, only Sulfadoxine-pyrimethamine (SP) and Sulfadoxine-pyrimethamine plus amodiaquine (SPAQ) are currently recommended by WHO for chemoprevention, which use is currently threatened by increasing resistance to SP. The strategy of the study sponsor, Medicines for Malaria Venture (MMV) is to re-combine existing and approved antimalarials used individually for the treatment of malaria, for the purpose of malaria chemoprevention. As part of this strategy, a review of the potential efficacy and duration of protection, the safety and tolerability, as well as the risk of emergence of resistance of currently approved products has been conducted, with a view to identify a new combination of two registered products that may be suitable for malaria chemoprevention.

A combination of pyronaridine tetraphosphate (PYR) and piperaquine tetraphosphate (PQP) was considered to have potential for this purpose. In the European Union, PQP is marketed in a fixed dose combination with the short acting antimalarial dihydroartemisinin (DHA) as Eurartesim® for treatment of acute uncomplicated malaria. PYR in a fixed dose combination with artesunate (AS) received positive scientific opinion from EMA through Article 58 and is marketed in South Korea and in many malaria endemic countries in Africa and South-East Asia as Pyramax® for treatment of acute uncomplicated malaria. The efficacy of both PYR and PQP combined to the artemisinin derivatives have been demonstrated in the treatment of uncomplicated malaria in various clinical trials in different regions and these combinations have been in clinical use for at least 20 and 40 years, respectively.

This study in healthy adults will be the first one to evaluate combined administration of pyronaridine tetraphosphate (PYR) and piperaquine tetraphosphate (PQP) in humans. A parallel group design (n=40) including a placebo cohort will be used to evaluate safety/tolerability and PK of the two treatments either as monotherapy or in combination. To our knowledge, this study will be the first human study with this new combination. The approved adult malaria treatment doses of PQP and PYR have been chosen for this trial and four treatment arms that include the use of matched placebos will facilitate discrimination of the contribution of the treatments to any safety/tolerability signal and determine the pharmacokinetic of PYR and PQP when administered alone and in combination.

Given the ultimate target population, the study will be carried out in healthy black participants of sub-Saharan African origin (defined as participants whose biological parents are both black and are of sub-Saharan African origin).

ELIGIBILITY:
Inclusion Criteria:

1. Black male or female, of Sub-Saharan African origin (defined as participants whose parents are both black and are of Sub-Saharan African origin) aged ≥18 years to ≤45 years at the date of signing informed consent. This inclusion criterion will only be assessed at the screening visit
2. Healthy as defined by:

   * the absence of clinically significant illness and surgery within four weeks prior to dosing. Participants vomiting within 24 hours pre-dose will be carefully evaluated for upcoming illness/disease. Inclusion pre-dosing is at the discretion of the Investigator
   * the absence of clinically significant history of neurological, endocrine, cardiovascular, respiratory, haematological, immunological, psychiatric, gastrointestinal, renal, hepatic and metabolic disease
3. Participants must agree to use the following contraceptive requirements for the applicable duration:

   * Female participants of non-childbearing potential (WNCBP): Defined as either postmenopausal (evidence of menopause based on a combination of amenorrhea for at least one year and increased serum follicle-stimulating hormone (FSH) level [>30 IU/L]), or surgical sterilisation (evidence of hysterectomy and/or bilateral oophorectomy) CONTRACEPTION REQUIRED: None
   * Female participants of childbearing potential (WOCBP) who anticipate being sexually active with a male during the trial (from one complete menstrual cycle prior to the first IMP administration until 13 weeks after the last IMP administration):

   CONTRACEPTION REQUIRED: Highly effective contraception must start one complete menstrual cycle prior to the first day of dosing and continue until 13 weeks after the last IMP administration. Highly effective contraception methods for WOCBP include:
   * combined (i.e. oestrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation:

     * oral
     * intravaginal
     * transdermal
   * progestogen-only hormonal contraception associated with inhibition of ovulation:

     * oral
     * injectable
     * implantable
   * intrauterine hormone-releasing system (IUS)
   * intrauterine device (IUD)
   * bilateral tubal occlusion
   * infertile male partner (e.g. vasectomised, permanently sterile following bilateral orchidectomy, or any other documented cause of infertility)
   * Female participants of childbearing potential (WOCBP) who agree to remain abstinent for the duration of the trial (from one complete menstrual cycle prior to the first IMP administration until 13 weeks after the last IMP administration):

   CONTRACEPTION REQUIRED: Abstinence (sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the trial treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant. Calendar, symptothermal and post-ovulation methods of contraception are not considered to be equivalent to abstinence)

   • Male participants, who agree to remain abstinent for the duration of the trial (from first IMP administration until 13 weeks after the last IMP administration): CONTRACEPTION REQUIRED: Abstinence (sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the trial treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the participant) If the situation changes post-dose during the trial, participants must use a condom with or without spermicide.

   • Male participants, who anticipate being sexually active during the trial period (from first IMP administration until 13 weeks after the last IMP administration) with a woman who is either a WOCBP, a woman who is pregnant and/or breast feeding:

   CONTRACEPTION REQUIRED: From the first day of dosing until the end of the systemic exposure of the trial drug. Acceptable methods are:
   * male condom with or without spermicide
   * infertile male (e.g. vasectomised, permanently sterile following bilateral orchidectomy, or any other documented cause of infertility)
4. Participants must agree not to donate sperm or ova from the time of the first administration of trial medication until three months after the end of the systemic exposure of the trial drug
5. Participants must have a body weight of 50 kg or greater and a BMI between 18.0 kg/m² - 28.0 kg/m² (inclusive) at screening
6. Satisfactory medical assessment with no clinically significant or relevant abnormalities as determined by medical history, physical examination, vital signs, 12-lead ECG and clinical laboratory evaluation (haematology, biochemistry, coagulation, and urinalysis) that is reasonably likely to interfere with the participant's participation in or ability to complete the trial as assessed by the Investigator
7. Ability to provide written, personally signed, and dated informed consent to participate in the trial, in accordance with the ICH Good Clinical Practice (GCP) Guideline E6 (R2) (2016) and applicable regulations, before completing any trial-related procedures
8. An understanding, ability, and willingness to fully comply with trial procedures and restrictions.

Exclusion Criteria:

1. Current or recurrent disease (e.g. cardiovascular, haematological, neurological, endocrine, immunological, renal, hepatic or gastrointestinal or other conditions, including cholecystectomy or gastrectomy) that could affect the action, absorption, distribution, metabolism or excretion of PYR or PQP or could affect clinical assessments or clinical laboratory evaluations
2. Any history of seizures or epilepsy
3. Any history of photosensitivity
4. Any documented retinopathy
5. History of malaria in the previous two years
6. A score of 20 or more on the Beck Depression Inventory, and/or a response of 1, 2 or 3 for item 9 of this inventory (related to suicidal ideation) [26].
7. Current or relevant history of physical or psychiatric illness that are not stable or may require a change in treatment, or use of prohibited therapies during the trial, that make the participant unlikely to fully comply with the requirements of the trial or to complete the trial, or any condition that presents undue risk from the investigational product or trial procedures
8. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participant at risk because of participation in the trial, or may influence the result of the trial or the participant's ability to participate in the trial
9. The history or presence of any of the following cardiac conditions: known structural cardiac abnormalities; family history of long QT syndrome; cardiac syncope or recurrent, idiopathic syncope; exercise-related clinically significant cardiac events
10. Any clinically significant abnormalities in rhythm, conduction or morphology of resting ECG or clinically important abnormalities that may interfere with the interpretation of QTc interval changes. This includes participants with any of the following (at screening or Day -1):

    * sinus node dysfunction
    * clinically significant PR >220 msecs (PQ) interval prolongation
    * second- or third-degree atrioventricular (AV) block
    * sustained cardiac arrhythmia's including (but not limited to) atrial fibrillation or supraventricular tachycardia, or any symptomatic arrhythmia, with the exception of isolated extra-systoles
    * abnormal T-wave morphology which may impact on the QT/QTc assessment
    * QT interval corrected using the Fridericia's formula (QTcF) >450 ms (males and females)
    * any other ECG abnormalities in the standard 12-lead ECG and 24-hour 12 lead Holter ECG or an equivalent assessment which in the opinion of the Investigator will interfere with the ECG analysis Participants with borderline abnormalities may be included if the deviations do not pose a safety risk, and if agreed between the appointed cardiologist and the PI.
11. Has vital signs consistently outside of normal range at screening or Day -1. Acceptable normal range is as follows:

    * supine HR 40 - 100 bpm (after at least five minutes of supine rest)
    * supine blood pressure (after at least five minutes of supine rest):

      * systolic blood pressure: 90 - 140 mmHg
      * diastolic blood pressure: 40 - 90 mmHg
12. Has a positive test for Hepatitis B surface Antigen (HBsAg), Hepatitis C Antibody (HCV Ab), or Human Immunodeficiency Virus Antibody (HIV Ab) at screening
13. Has total bilirubin, ALT or AST consistently >ULN at screening (up to two repeats may be taken during the screening period; volunteer may be included if two out of the three total results are ≤ULN), or has total bilirubin, ALT or AST>ULN on Day -1 (mild variations from baseline may be allowed if considered not clinically significant by the Investigator)
14. Has a haemoglobin, platelet count, total white blood cell count, lymphocyte or monocyte count less than Lower Limit of Normal (LLN) (up to two repeats may be taken during the screening period and on Day -1 (participants may be included if two out of the three total results are greater or equal to LLN), at screening. Where there is a clear diurnal effect on the result participants may be included if variations are considered not clinically relevant by the Investigator
15. Any other abnormal findings on vital signs, ECG, physical examination or laboratory evaluation of blood and urine samples that the Investigator judges as likely to interfere with the trial or pose an additional risk in participating
16. Positive test results for alcohol or drugs of abuse at screening or Day -1
17. Female participants who are pregnant (including a positive serum pregnancy test at screening or on Day -1) or breastfeeding
18. Male participants with a female partner(s) who is (are) pregnant or lactating at screening or on Day -1, or is (are) expected to be during the trial period
19. History or clinical evidence of substance and/or alcohol abuse within the two years before screening. Alcohol abuse is defined as regular weekly intake of more than 14 units (for both males and females), using the following National Health Service (NHS) alcohol tracker https://www.nhs.uk/oneyou/for-your-body/drink-less/know-your-alcohol-units/
20. Treatment with an investigational drug within 90 days or five half-lives preceding the first dose of trial medication (whichever is the longer)
21. Use of tobacco in any form (e.g. smoking or chewing) or other nicotine-containing products in any form (e.g. gum, patch, electronic cigarettes) within six months prior to the planned first day of dosing
22. Has used any medication (see list for reference: https://www.fda.gov/drugs/drug-interactions-labeling/drug-development-and-drug-interactions-table-substrates-inhibitors-and-inducers#transporter ) that is either a moderate or strong inhibitor or inducer of CYP3A4 within 30 days or five half-lives (whichever is longer) prior to the planned first day of dosing
23. Additionally, participants must have not consumed other substances known to be potent inhibitors or inducers of CYP3A4 system such as grapefruit or cranberry juice-containing products in the 30 days before the planned first IMP administration
24. Has used any other prescription medication (excluding hormonal contraception and hormone replacement therapy) within 14 days or five half-lives (whichever is longer) prior to Day 1 of the dosing period that the Investigator judges is likely to interfere with the trial or pose an additional risk in participating
25. Has used any over-the-counter medication (including multivitamin, herbal, or homeopathic preparations;) during the seven days or five half-lives of the medication (whichever is longer) prior to Day 1 of the dosing period, that the Investigator judges is likely to interfere with the trial or pose an additional risk in participating
26. Consumption of any herbal remedies or dietary supplements containing a herbal remedy in the 30 days before the planned Day 1 of the dosing period
27. Ingestion of any poppy seeds within the 24 hours prior to screening and admission
28. Known or suspected intolerance or hypersensitivity to the investigational products, any closely related compound, or any of the stated ingredients
29. History of significant allergic reaction (e.g. anaphylaxis, angioedema, but excluding untreated, asymptomatic, seasonal allergies) to any product (food, pharmaceutical, etc)
30. Donation of blood or blood products (excluding plasma) within 90 days prior to trial medication administration
31. Has a mental incapacity or language barriers precluding adequate understanding, co-operation, or compliance with the trial requirements
32. An inability to follow a standardised diet and meal schedule or inability to fast, as required during the trial
33. Inability to swallow eight tablets in short succession
34. Participants with veins on either arm that are unsuitable for intravenous puncture or cannulation (e.g. veins that are difficult to locate, or a tendency to rupture during puncture)
35. Prior screen failure (where the cause of the screen failure is not deemed to be temporary), randomisation, participation, or enrolment in this trial. Participants who initially failed due to temporary non-medically significant issues are eligible for re-screening once the cause has resolved
36. Participants who have received or are planning on receiving a COVID-19 vaccination four weeks before first dose administration, or within one week after trial completion
37. Any conditions which in the opinion of the Investigator would make the volunteer unsuitable for enrolment or could interfere with the participants' participation in or completion of the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Chalon, MD PhD, Study Director — MMV Medicines for Malaria Venture; Ulrike Lorch, MD, Principal Investigator — Richmond Pharmacology Limited
Locations (1):
- Richmond Pharmacology Ltd, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Felices M, Borghini-Fuhrer I, Abla N, Chalon S. Concentration-Response Analysis of the Combination of Pyronaridine and Piperaquine on Corrected QT Interval From a Randomized, Double-Blind, Placebo-Controlled Study in Healthy Adults of African Sub-Saharan Origin. Clin Transl Sci. 2025 Jul;18(7):e70305. doi: 10.1111/cts.70305. PMID 40689586

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 37 participants of the expected 40 participants were enrolled at a Phase 1 Pharmacology Unit in London, UK. The first volunteer was enrolled on 14Feb2022. A total of 87 volunteers were screened, ultimately 37 participants were dosed.
Period: Overall Study
Arm/Group | PYR and PQP Combination | PYR and Placebo Combination | PQP and Placebo Combination | Placebo Combination
Started | 15 | 8 | 8 | 6
Completed | 15 | 8 | 8 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Sponsor and Investigator decision to halt recruitment when 37 of the expected 40 participants had been dosed.
Groups:
- Total: Total of all reporting groups
Arm/Group | PYR and PQP Combination | PYR and Placebo Combination | PQP and Placebo Combination | Placebo Combination | Total
Number analyzed (Participants) | 15 | 8 | 8 | 6 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 15 | 8 | 8 | 6 | 37
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: Years] | 27 [18 to 36] | 30.5 [21 to 38] | 27.9 [21 to 38] | 26 [19 to 35] | 27.8 [18 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 5 | 4 | 21
  Male | 7 | 4 | 3 | 2 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Sub-Saharan African origin | 15 | 8 | 8 | 6 | 37
Region of Enrollment [Number; unit: participants]
  United Kingdom | 15 | 8 | 8 | 6 | 37

OUTCOME MEASURES:

1. Primary Outcome: The Incidence, Severity and Relationship of Treatment-Emergent Adverse Events (TEAEs).
Time Frame: From start of IP administration - to follow up visit, Day 30
Population: Participants
Measure: Number; unit: participants
Arm/Group | PYR and PQP Combination | PYR and Placebo Combination | PQP and Placebo Combination | Placebo Combination
Number analyzed (Participants) | 15 | 8 | 8 | 6
participants
  number of participants with at least one TEAE | 10 | 7 | 4 | 5
  number of participants with at least one Related TEAE | 5 | 5 | 2 | 0
  number of participants with at least one Mild TEAE | 9 | 6 | 4 | 5
  number of participants with at least one Moderate TEAE | 2 | 0 | 0 | 0
  number of participants with at least one Severe TEAE | 2 | 2 | 0 | 0

ADVERSE EVENTS:
Time Frame: From start of IP administration to follow-up visit at Day 30
Arm/Group | PYR and PQP Combination | PYR and Placebo Combination | PQP and Placebo Combination | Placebo Combination
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/8 | 0/8 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/8 | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 10/15 | 7/8 | 4/8 | 5/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PYR and PQP Combination (N=15) | PYR and Placebo Combination (N=8) | PQP and Placebo Combination (N=8) | Placebo Combination (N=6)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postural Dizziness (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual Impairment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Change of Bowel Habit (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Frequent Bowel Movements (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Systemic Viral Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Musculokeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the Sponsor and RPL agree that it will be desirable to publish the results of this trial; both parties will liaise in good faith to publish the results. RPL agree to obtain the Sponsor's prior written approval of such publications.

DOCUMENTS (3):
  • Study Protocol (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT05160363/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-17): https://cdn.clinicaltrials.gov/large-docs/63/NCT05160363/SAP_001.pdf
  • Informed Consent Form (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT05160363/ICF_002.pdf